CLINICAL TRIAL: NCT04338412
Title: Evaluating Optimal Operating Table Height for ProSeal-LMA™ Insertion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Azlina Masdar, Dr, National University of Malaysia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Other
Other Study IDs: AzlinaM
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Evaluation of Optimal Operating Table Height for Successful Placement of Proseal Laryngeal Mask Airway
Keywords: Proseal LMA; Table height; LMA placement; Body landmark

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group U (Active Comparator): Performers' umbilicus
  Interventions: Device: ProSeal-LMA™
- Group R (Active Comparator): Performers' lowest rib margin
  Interventions: Device: ProSeal-LMA™
- Group X (Active Comparator): Performers' xiphoid process
  Interventions: Device: ProSeal-LMA™

INTERVENTIONS:
Device: ProSeal-LMA™ — It is a second generation LMA that is commonly used among all other LMAs

SUMMARY:
Usage of LMA has gained much importance especially as a rescue device for failed intubation. We hypothesised optimal operating table height could improve successful attempt of ProSeal-LMA™ (P-LMA™) insertion.

The main objective of this study is to evaluate the optimal operating table height for successful placement of P-LMA™ by comparing operating table height to operators' body landmark.

The secondary objectives of this study are to evaluate duration required for a successful P-LMA™ insertion and its associated complications during the attempt.

DETAILED DESCRIPTION:
Written informed consent will be obtained by primary investigator from patients recruited into this study. The study will be conducted by anesthesiology medical officers with more than 3 years of anesthetic experience.

All recruited patients will be reviewed by the primary investigator prior to their operation. Patients' demographic characteristics and airway assessment will be recorded preoperatively. Airway assessment consists of Mallampati score, mouth opening and thyromental distance (TMD). Mallampati score is assessed based on modified Samsoon and Young test. Mouth opening is taken as distance between upper and lower incisor teeth when mouth is maximally opened. TMD is measured as distance between symphysis menti and thyroid notch with the head in full extension. Patients are required to be fasted for at least 6 hours before the scheduled operation. They will then be randomly allocated by computer generated randomisation into one of three groups based on height of operating table with reference to the performers' anatomical landmark. The height of the operating table will be adjusted at levels corresponding to the performers' umbilicus (Group U), lowest rib margin (Group R) or xiphoid process (Group X).

In the operation theatre, standard monitoring will be applied. Operating table will be adjusted according to the respective group randomization. Patient will be preoxygenated with 100% oxygen until end-tidal oxygen (etO2) of 85% is achieved. Following which, intravenous (IV) anesthetic induction drugs will be given: fentanyl 1.5 mcg/kg, propofol 2.0 mg/kg. After loss of consciousness, the attending anesthesiology medical officer will proceed with mask ventilation with a mixture of oxygen and sevoflurane to achieve Minimum Alveolar Concentration (MAC) of 1.0 to 1.2. If there is no difficult ventilation, IV rocuronium 0.6 mg/kg will be given and the patient will be subsequently ventilated for 3 minutes. If unexpected difficult ventilation occurs, patient will be drop out from this study and management of the patient will be at the discretion of attending anesthesiologist.

P-LAM™ will then be inserted by the attending anesthesiology medical officer. The size of P-LMA™ used will be according to the manufacturer's recommendation. The P-LMA™ will be thoroughly checked and tested as per manufacturer recommendations i.e.: visual inspection and; inflation and deflation test. All P-LMA™ are reuse within the manufacturers' recommendation, i.e. ≤40 usages and manufactured by The Laryngeal Mask Airway Co Ltd, Mahe, Seychelles.

The P-LMA™ will be inserted with cuff fully deflated using introducer technique on all attempts. Patient's head will be positioned with flexion of the neck and extension of the head using operator's non-dominant hand. The P-LMA™ is held and inserted while pressing up against palate and posterior pharyngeal wall until resistance is felt. P-LMA™ cuff is inflated with a volume of air recommended by the manufacturer. The P-LMA™ cuff pressure is then measured by a cuff pressure manometer to ensure cuff pressure achieves 60 cmH2O.

A successful insertion is determined when it fulfills both positional and performance tests. Positional tests includes gastric tube 'bubble' test, suprasternal notch tap test and insertion of gastric tube through its drain tube which verifies the ideal position of P-LMA™ placement. Another set of test known as performance test consists of oropharyngeal leak pressure test and it determines how well P-LMA™ is able to perform once it is inserted. All these tests will be done after insertion and are recorded by a second anesthesiology medical officer who was not involved in the insertion process. General anesthesia is maintained with a mixture of oxygen/air (50%/50%) and sevoflurane to achieve Minimum Alveolar Concentration (MAC) of 1.0 to 1.2 intraoperatively.

Gastric tube 'bubble' test is done by sealing the drainage tube of P-LMA™ with a drop of gel 2-3 mm height followed by Intermittent Positive Pressure Ventilation (IPPV) with a tidal volume of 8 ml/kg. If no air leak out and gel remains in the drainage tube, it suggests good P-LMA™ placement. Suprasternal notch test is done by placing a drop of gel 2-3 mm height and a firm pressure is applied to suprasternal notch with a finger. P-LMA™ placement is considered good if gel column moves synchronously with the applied pressure. Successful insertion of a 14 Fr or 16 Fr orogastric tube via drainage tube without encountering any resistance and confirmation of its position in gastric suggests a good P-LMA™ placement. Position of orogastric tube is verified by presence of gastric fluid aspiration and audible gastric insufflation at the epigastrium during auscultation via stethoscope after 20 ml injection of air.

Subsequently, to test for oropharyngeal leak pressure test, airway seal pressure is determined by setting Adjustable Pressure Limiting (APL) valve to 30 cmH2O and fresh gas flow at ≥3 L/min. A good oropharyngeal leak pressure is determined by its capability to record a stable airway pressure of ≥25 cmH2O in supine position and such recording suggests a good P-LMA™placement.

The same assistant who records the data will also record duration taken for P-LMA™ insertion by using a standard stopwatch and it starts from the time when operator places the P-LMA™ at the aperture of oral orifice till appearance of first end-tidal CO2 (etCO2) waveform on capnography. Time measurement is only done during the first P-LMA™insertion.

If there is a failure of insertion or failure of placement of P-LMA™ during the first attempt, defines as any failure of individual positional and performance tests, the patient will be considered as failed P-LMA™ attempt and subsequently airway management will be up to the discretion of the attending anesthesiologist. Ease of placement of P-LMA™ is evaluated by the operator via subjective ease of insertion whereby score 1=very easy, 2=easy, 3=difficult, 4=very difficult. Presence of airway morbidity during the first attempt of P-LMA™ insertion will be recorded. Examples of complications monitored includes oxygen desaturation of <90%, airway obstruction, laryngospasm, bronchospasm and oropharyngeal trauma (defined as presence of blood upon removal of P-LMA™). After the procedure is done, operating table height will be adjusted according to surgical operation requirements.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 65 years old
2. American Society of Anesthesiologists (ASA) I-II patients
3. Elective and emergency surgeries requiring general anaesthesia where use of P-LMA™ is not contraindicated

Exclusion Criteria:

1. Congenital or acquired airway abnormality
2. Cervical spine pathology
3. Edentulous or loose tooth
4. BMI ≥35 kg/m2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Optimal operating table height for successful placement of P-LMA™ | 2 years
  To evaluate optimal operating table height for successful placement of P-LMA™ by comparing operating table height to operators' body landmark

SECONDARY OUTCOMES:
Evaluation of time required for a successful P-LMA™ insertion | 2 years
  To evaluate duration of time required for a successful P-LMA™ insertion and its associated complications during the attempt
Evaluation of associated complications during P-LMA™ insertion | 2 years
  To evaluate associated complications during P-LMA™ insertion

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Kebangsaan Malaysia Medical Centre, Kuala Lumpur, Malaysia